CLINICAL TRIAL: NCT04156451
Title: Effectiveness of Fluid Deresuscitation With Central Venous Pressure Target 0-4 mmHg on Capillary Perfusion Density, Acute Kidney Injury Stage, Cardiac Index, and the Intensive Care Unit Length of Stay in Septic Shock Patients After Resuscitation
Brief Title: Effect of Fluid Deresuscitation With Central Venous Pressure Target 0-4 mmHg in Septic Shock Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Dita Aditianingsih, MD, PhD, Anesthesiologist Consultant, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IndonesiaUAnes040
Record Dates: First submitted 2019-11-01; First posted 2019-11-07 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Septic Shock
Keywords: Deresuscitation; Central Venous Pressure; Septic Shock; Furosemide
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Central Venous Pressure 8 - 10 mmHg (Active Comparator): Furosemide deresuscitation or crystalloid loading until the CVP target 8-12 mmHg is reached
  Interventions: Procedure: Fluid resuscitation and furosemide administration (bolus and continuous) with central venous pressure target 8 - 10 mmHg
- Central Venous Pressure 0 - 4 mmHg (Experimental): Furosemide deresuscitation or crystalloid loading until the CVP target 0-4 mmHg is reached
  Interventions: Procedure: Fluid deresuscitation and furosemide administration (bolus and continuous) with central venous pressure target 0 - 4 mmHg

INTERVENTIONS:
Procedure: Fluid resuscitation and furosemide administration (bolus and continuous) with central venous pressure target 8 - 10 mmHg — Crystalloid loading or furosemide administration with the CVP target 8-10 mmHg is reached in septic shock patients
  Arms: Central Venous Pressure 8 - 10 mmHg
Procedure: Fluid deresuscitation and furosemide administration (bolus and continuous) with central venous pressure target 0 - 4 mmHg — active fluid removal with furosemide bolus and continuous or crystalloid loading until the CVP target 0-4 mmHg is reached in septic shock patients
  Arms: Central Venous Pressure 0 - 4 mmHg

SUMMARY:
A scientific research to prove the safety and effectiveness of TVS 0 - 4 mmHg as a target of resuscitation using furosemide, to improve Perfused Vessel Density (PVD) > 25 mm / mm2, AKI stage (based on KDIGO criteria), CI > 2.5 cc / min / m2 , prevent the incidence of intubation, reduce the duration of ventilator use <120 hours and reduce the length of ICU stay in patients with septic shock after resuscitation

DETAILED DESCRIPTION:
The study aims to evaluate the effectiveness of deresuscitation with target CVP 0 - 4 mmHg on septic shock patients in the ICU on capillary perfusion density, AKI stage (based on KDIGO criteria), the incidence of intubation, duration of use of mechanical ventilation, and length of stay in the ICU which can reduce the number of morbidity and mortality.

The study evaluates the difference in capillary perfusion density, AKI stage (based on KDIGO criteria), and the Cardiac index value between groups septic shock patients with CVP 0-4 mmHg on the 7th day after deresuscitation compared with the control group (CVP 8-10 mmHg on the first 7th day after being given deresuscitation).

The study evaluates the difference in the number of intubation incidents, duration of use ventilators, and care in the ICU between groups of patients with septic shock CVP 0 - 4 on day 28 after being given a degree of comparison with a control group (CVP 8-10 mmHg on day 28th after being deresuscitation).

ELIGIBILITY:
Inclusion Criteria:

* Septic shock patients who meet the diagnosis criteria for quick SOFA and KDIGO 1 stage AKI (creatinine value 1.5 times OR creatinine value> 0.3 initial OR urine production <0.5 ml/kg/hour for 6-12 hours
* Patients, both men and women, in the age range of 18 - 60 years
* Patients who experience post clean operative sepsis
* Patients who agree to attend the study by signing informed consent

Exclusion Criteria:

* Patients with primary heart problems, right or heart failure suffer from congenital heart disease
* Have severe chronic obstructive pulmonary disease, patients with severe pleural effusion
* Patients who, based on ultrasound examination, found stones or tumors in the kidney during the study period
* CKD patients are based on history taking and physical examination
* DNR (do not resuscitate) patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Capillary Perfusion Density | 7 days
  Capillary Perfusion Density measurement using MicroScan every 24 hours during deresuscitation

SECONDARY OUTCOMES:
Acute Kidney Injury Stage | 7 days
  AKI staging using KDIGO criteria every 24 hours during deresuscitation
Cardiac Index | 7 days
  cardiac index measurement using bio-impedance cardiometry every 24 hours during deresuscitation
Neutrophil Gelatinase-Associated lipocalin (NGAL) | 1st and 7th day
  NGAL measurement from urinary sample using NGAL ELISA method at 1st and 7th day during deresuscitation
Renal Resistive Index (RRI) | 1st and 7th day
  RRI measurement using renal doppler ultrasonography at 1st and 7th day during deresuscitation
Length of ICU stay | 28 days
  length of ICU stay in days during and after deresuscitation

CONTACTS AND LOCATIONS:
Locations (1):
- Rumah Sakit Cipto Mangunkusumo, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vincent JL, Sakr Y, Sprung CL, Ranieri VM, Reinhart K, Gerlach H, Moreno R, Carlet J, Le Gall JR, Payen D; Sepsis Occurrence in Acutely Ill Patients Investigators. Sepsis in European intensive care units: results of the SOAP study. Crit Care Med. 2006 Feb;34(2):344-53. doi: 10.1097/01.ccm.0000194725.48928.3a. PMID 16424713
- [Background] Opal SM, Laterre PF, Francois B, LaRosa SP, Angus DC, Mira JP, Wittebole X, Dugernier T, Perrotin D, Tidswell M, Jauregui L, Krell K, Pachl J, Takahashi T, Peckelsen C, Cordasco E, Chang CS, Oeyen S, Aikawa N, Maruyama T, Schein R, Kalil AC, Van Nuffelen M, Lynn M, Rossignol DP, Gogate J, Roberts MB, Wheeler JL, Vincent JL; ACCESS Study Group. Effect of eritoran, an antagonist of MD2-TLR4, on mortality in patients with severe sepsis: the ACCESS randomized trial. JAMA. 2013 Mar 20;309(11):1154-62. doi: 10.1001/jama.2013.2194. PMID 23512062
- [Background] Dellinger RP, Levy MM, Carlet JM, Bion J, Parker MM, Jaeschke R, Reinhart K, Angus DC, Brun-Buisson C, Beale R, Calandra T, Dhainaut JF, Gerlach H, Harvey M, Marini JJ, Marshall J, Ranieri M, Ramsay G, Sevransky J, Thompson BT, Townsend S, Vender JS, Zimmerman JL, Vincent JL; International Surviving Sepsis Campaign Guidelines Committee; American Association of Critical-Care Nurses; American College of Chest Physicians; American College of Emergency Physicians; Canadian Critical Care Society; European Society of Clinical Microbiology and Infectious Diseases; European Society of Intensive Care Medicine; European Respiratory Society; International Sepsis Forum; Japanese Association for Acute Medicine; Japanese Society of Intensive Care Medicine; Society of Critical Care Medicine; Society of Hospital Medicine; Surgical Infection Society; World Federation of Societies of Intensive and Critical Care Medicine. Surviving Sepsis Campaign: international guidelines for management of severe sepsis and septic shock: 2008. Crit Care Med. 2008 Jan;36(1):296-327. doi: 10.1097/01.CCM.0000298158.12101.41. PMID 18158437
- [Background] Dellinger RP, Levy MM, Rhodes A, Annane D, Gerlach H, Opal SM, Sevransky JE, Sprung CL, Douglas IS, Jaeschke R, Osborn TM, Nunnally ME, Townsend SR, Reinhart K, Kleinpell RM, Angus DC, Deutschman CS, Machado FR, Rubenfeld GD, Webb SA, Beale RJ, Vincent JL, Moreno R; Surviving Sepsis Campaign Guidelines Committee including the Pediatric Subgroup. Surviving sepsis campaign: international guidelines for management of severe sepsis and septic shock: 2012. Crit Care Med. 2013 Feb;41(2):580-637. doi: 10.1097/CCM.0b013e31827e83af. PMID 23353941
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Prowle JR, Echeverri JE, Ligabo EV, Ronco C, Bellomo R. Fluid balance and acute kidney injury. Nat Rev Nephrol. 2010 Feb;6(2):107-15. doi: 10.1038/nrneph.2009.213. Epub 2009 Dec 22. PMID 20027192
- [Background] Payen D, de Pont AC, Sakr Y, Spies C, Reinhart K, Vincent JL; Sepsis Occurrence in Acutely Ill Patients (SOAP) Investigators. A positive fluid balance is associated with a worse outcome in patients with acute renal failure. Crit Care. 2008;12(3):R74. doi: 10.1186/cc6916. Epub 2008 Jun 4. PMID 18533029
- [Background] Van Biesen W, Yegenaga I, Vanholder R, Verbeke F, Hoste E, Colardyn F, Lameire N. Relationship between fluid status and its management on acute renal failure (ARF) in intensive care unit (ICU) patients with sepsis: a prospective analysis. J Nephrol. 2005 Jan-Feb;18(1):54-60. PMID 15772923
- [Background] Wang CH, Hsieh WH, Chou HC, Huang YS, Shen JH, Yeo YH, Chang HE, Chen SC, Lee CC. Liberal versus restricted fluid resuscitation strategies in trauma patients: a systematic review and meta-analysis of randomized controlled trials and observational studies*. Crit Care Med. 2014 Apr;42(4):954-61. doi: 10.1097/CCM.0000000000000050. PMID 24335443
- [Background] Cordemans C, De Laet I, Van Regenmortel N, Schoonheydt K, Dits H, Huber W, Malbrain ML. Fluid management in critically ill patients: the role of extravascular lung water, abdominal hypertension, capillary leak, and fluid balance. Ann Intensive Care. 2012 Jul 5;2(Suppl 1 Diagnosis and management of intra-abdominal hyperten):S1. doi: 10.1186/2110-5820-2-S1-S1. eCollection 2012. PMID 22873410